CLINICAL TRIAL: NCT01873365
Title: Physician-practice Based Cohort Study to Estimate the Burden of Herpes Zoster and Postherpetic Neuralgia in Japan
Brief Title: A Study to Assess the Burden of Herpes Zoster and Postherpetic Neuralgia in Japanese Adults Aged Sixty Years and Above
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 200089
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Herpes Zoster
Keywords: Quality of life; Herpes zoster; Postherpetic neuralgia; Japan; Physician-practice; Adults; Health economics
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prospective Group: Japanese adults, aged greater than or equal to sixty years, diagnosed with HZ.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Case report forms (CRFs), logbooks and booklets.

SUMMARY:
The study aims to estimate the incidence of herpes zoster (HZ), proportion of postherpetic neuralgia (PHN) and the economic burden and impact on quality of life, in Japanese adults greater than or equal to sixty years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* A male or female greater than or equal to sixty years of age, presenting with HZ at the time of enrollment.
* HZ diagnosis.

  * Is the subject's first outpatient diagnosis for this HZ episode. OR
  * Took place up to seven days prior to the initial visit for the present study. Note: Recurrent HZ cases may be enrolled as new cases based on the investigator's clinical practice.

Exclusion Criteria:

• Not applicable.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese adults, male or female, greater than or equal to sixty years of age, presenting with HZ at the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2013-06-29; Primary Completion 2015-02-04 (Actual); Study Completion 2015-02-04 (Actual)

PRIMARY OUTCOMES:
Total number of HZ cases reported in the study area, overall and within a specific age-group and gender. The following age-groups will be considered: 60-69, 70-79 and ≥ 80 years of age. | Approximately 1 year
Occurrence of HZ-associated PHN pain, persisting between 90 and 270 days after the initial visit for this study. | Day 90 - Day 270

SECONDARY OUTCOMES:
Occurrence of HZ-associated hospitalisations. | Day 0 - Day 270
Occurrence of HZ-associated any pain, persisting between 0 and 270 days after the initial visit for this study. | Day 0 - Day 270
Anamnestic information, clinical parameters and complications related to HZ. | Day 0 - Day 270
Direct medical, direct non-medical and indirect costs related to HZ. | Day 0 - Day 90
Quality of life (QoL) assessment in HZ subjects. | Day 0 - Day 90
Direct medical, direct non-medical and indirect costs related to PHN. | Day 90 - Day 270
QoL assessment in PHN subjects. | Day 90 - Day 270
Impact of the following factors on the development of PHN: - age, - gender, - concomitant disease, - current immunosuppressive therapy, - HZ severity at first consultation, - timing of initiation of treatment with antiviral agent etc. | Day 0 - Day 270

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hokkaido, Japan

REFERENCES:
- [Derived] Mizukami A, Sato K, Adachi K, Matthews S, Holl K, Matsuki T, Kaise T, Curran D. Impact of Herpes Zoster and Post-Herpetic Neuralgia on Health-Related Quality of Life in Japanese Adults Aged 60 Years or Older: Results from a Prospective, Observational Cohort Study. Clin Drug Investig. 2018 Jan;38(1):29-37. doi: 10.1007/s40261-017-0581-5. PMID 29086340
- [Derived] Nakamura H, Mizukami A, Adachi K, Matthews S, Holl K, Asano K, Watanabe A, Adachi R, Kiuchi M, Kobayashi K, Sato K, Matsuki T, Kaise T, Curran D. Economic Burden of Herpes Zoster and Post-Herpetic Neuralgia in Adults 60 Years of Age or Older: Results from a Prospective, Physician Practice-Based Cohort Study in Kushiro, Japan. Drugs Real World Outcomes. 2017 Dec;4(4):187-198. doi: 10.1007/s40801-017-0119-4. PMID 28988331
- [Derived] Sato K, Adachi K, Nakamura H, Asano K, Watanabe A, Adachi R, Kiuchi M, Kobayashi K, Matsuki T, Kaise T, Gopala K, Holl K. Burden of herpes zoster and postherpetic neuralgia in Japanese adults 60 years of age or older: Results from an observational, prospective, physician practice-based cohort study. J Dermatol. 2017 Apr;44(4):414-422. doi: 10.1111/1346-8138.13639. Epub 2016 Dec 5. PMID 27917531